CLINICAL TRIAL: NCT05730244
Title: A Single Arm No-treatment Self-controlled Trial Pilot Study Evaluating the Clinical Efficacy and Safety Profile of 20% Cassia Alata Cream Against Tinea Versicolor
Brief Title: A Study of the Clinical Efficacy and Safety of 20% Cassia Alata Extract Against Tinea Versicolor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC-MN.29, 2021/2022
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Tinea Versicolor; Pityriasis Versicolor
Keywords: Tinea Versicolor,; Cassia alata extract; Pityriasis versicolor
MeSH Terms: conditions — Tinea Versicolor

STUDY DESIGN:
Intervention Model Description: A self-controlled trial pilot study evaluating the clinical efficacy and safety profile of 20% Cassia alata cream against tinea versicolor.
  Single group, all with tinea versicolor. Selected area treated, untreated areas serve as internal control. Assessment using background spontaneous clearance data and internal control comparison from non-treated areas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants with tinea versicolor who will have a treatment site selected. We will leave untreated areas to serve as "internal controls". Participants will apply cream to the designated areas but leave non-designated untreated. At follow up visits we will do fungal scrapings, visual examination and Wood's lamp evaluation of treatment and non-treatment areas
  Interventions: Drug: 20% Cassia alata cream

INTERVENTIONS:
Drug: 20% Cassia alata cream — Thin layer of cassia alata cream to cover treatment area. 1 finger tip unit will cover roughly 4 x 4 inch area. Number of FTU determined by investigators depending on rough size of area to be treated

SUMMARY:
The goal of this clinical trial is to establish the efficacy of Cassia alata extract as a cream form in treating tinea versicolor (liver spots/shifting clouds). The main questions the study aims to answer are:• Does the use of this extract help resolve tinea versicolor better than no treatment? Does the use of this cream have significant side effects i.e, is it safe? Participants will be asked to treat a designated area while leaving additional areas untreated. 1-2 finger tip units of cream will be applied to the treatment site twice daily at least 8 hours apart. Participants will attend the trial clinic every 4 weeks for 12 weeks.

DETAILED DESCRIPTION:
Tinea (pityriasis) versicolor is a common superficial fungal infection. A variety of topical antifungals are used in its treatment. In Jamaica, many people use crushed leaves of the Cassia alata plant (Senna alata) as a traditional remedy. Rare investigators have described its activity against the causative fungus, Malassezia spp. Aim: We wish to confirm the efficacy of the extract, devise dosing regimen, document potential side effects Study Design/Methodology: A single-arm arm no-treatment self-controlled trial pilot study evaluating the clinical efficacy and safety profile of 20% Cassia alata cream against tinea versicolor. Therapeutic efficacy reported as clinical and microbiological resolution of tinea versicolor in treated area will be assessed and compared with non-treated areas. Side effects and ease of use will be evaluated for and reported. Assessment will occur at baseline, 1 week, 4 weeks, 8 weeks and 12 weeks. Demographics will be tabulated and categorical variables generated. Associations of the presence/absence of these variables within both groups will be evaluated for using chi-squared tests. Results will be analyzed using SPSS version 26. Location: Dermatology Division (Room 13 Dept of Pathology) at University Hospital of the West Indies. Data Storage: Unique study ID, locked room and password protected computer belonging to the principal investigator. Only approved study investigators will have access. Time frame: 24 months months Confidentiality Statement: This study requires approval by the Ethics Committee, will require an informed consent and will comply with ethical rules governing research using human subjects, patient confidentiality and non-coercion as detailed within the proposal.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-89 of either sex
* Clinical features suggestive of tinea versicolor AND Microscopic confirmation using skin scraping stains with chlorazol black preparation AND/OR Wood's lamp fluorescence
* No treatment for versicolor in the preceding 4 weeks
* No contraindications to the application of C.alata cream including
* No history of allergy to C. alata
* No history of preservative allergy

Exclusion Criteria:

* Age <18 or >89 years
* Pregnant females
* History of hypersensitivity to C. alata or preservative
* Treatment within 4 weeks prior to enrollment
* Lesions which do not meet the diagnostic criteria of tinea versicolor

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Lesion Clearance | 12 weeks
  Proportion of participants with no visible lesions on which treatment applied. We will visually compare to baseline images and untreated skin
Fungal load | 12 weeks
  Change in the fungal load on skin scraping. We will looks for decrease in positivity and density in treated skin compared with baseline and untreated control skin

SECONDARY OUTCOMES:
Local skin reactions | 12 weeks
  Proportion of participants with new skin reactions (burning, pain, pruritus, blisters, color change)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Ho, MBBS, D.Sc, Principal Investigator — The University of the West Indies, Mona Campus
Locations (1):
- University of the West Indies, Mona, Kingston, Other, Jamaica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kallini JR, Riaz F, Khachemoune A. Tinea versicolor in dark-skinned individuals. Int J Dermatol. 2014 Feb;53(2):137-41. doi: 10.1111/ijd.12345. Epub 2013 Dec 10. PMID 24320140
- [Background] Gupta AK, Lyons DC. Pityriasis versicolor: an update on pharmacological treatment options. Expert Opin Pharmacother. 2014 Aug;15(12):1707-13. doi: 10.1517/14656566.2014.931373. Epub 2014 Jul 3. PMID 24991691
- [Background] Palanichamy S, Nagarajan S. Antifungal activity of Cassia alata leaf extract. J Ethnopharmacol. 1990 Jul;29(3):337-40. doi: 10.1016/0378-8741(90)90043-s. No abstract available. PMID 2214817
- [Background] Agarwal SK, Singh SS, Verma S, Kumar S. Antifungal activity of anthraquinone derivatives from Rheum emodi. J Ethnopharmacol. 2000 Sep;72(1-2):43-6. doi: 10.1016/s0378-8741(00)00195-1. PMID 10967452
- [Background] Barros Cota B, Batista Carneiro de Oliveira D, Carla Borges T, Cristina Catto A, Valverde Serafim C, Rogelis Aquiles Rodrigues A, Kohlhoff M, Leomar Zani C, Assuncao Andrade A. Antifungal activity of extracts and purified saponins from the rhizomes of Chamaecostus cuspidatus against Candida and Trichophyton species. J Appl Microbiol. 2021 Jan;130(1):61-75. doi: 10.1111/jam.14783. Epub 2020 Jul 29. PMID 32654270
- [Background] Zhang D, Fu Y, Yang J, Li XN, San MM, Oo TN, Wang Y, Yang X. Triterpenoids and Their Glycosides from Glinus Oppositifolius with Antifungal Activities against Microsporum Gypseum and Trichophyton Rubrum. Molecules. 2019 Jun 12;24(12):2206. doi: 10.3390/molecules24122206. PMID 31212847
- [Background] Damodaran S, Venkataraman S. A study on the therapeutic efficacy of Cassia alata, Linn. leaf extract against Pityriasis versicolor. J Ethnopharmacol. 1994 Mar;42(1):19-23. doi: 10.1016/0378-8741(94)90018-3. PMID 8046939
- [Background] Thamlikitkul V, Bunyapraphatsara N, Dechatiwongse T, Theerapong S, Chantrakul C, Thanaveerasuwan T, Nimitnon S, Boonroj P, Punkrut W, Gingsungneon V, et al. Randomized controlled trial of Cassia alata Linn. for constipation. J Med Assoc Thai. 1990 Apr;73(4):217-22. PMID 2203870
- [Background] Kaneko T, Makimura K, Onozaki M, Ueda K, Yamada Y, Nishiyama Y, Yamaguchi H. Vital growth factors of Malassezia species on modified CHROMagar Candida. Med Mycol. 2005 Dec;43(8):699-704. doi: 10.1080/13693780500130564. PMID 16422299